CLINICAL TRIAL: NCT07362628
Title: Ultrasound Guidance Versus Conventional Technique for Radial Arterial Puncture in Patients With Shock in the Emergency Department: A Randomized Controlled Trial
Brief Title: US Guidance for Radial Arterial Puncture in Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ismail Erkan Aydin (Other)
Responsible Party: Sponsor-Investigator, Ismail Erkan Aydin, Assistant Professor, Alanya Alaaddin Keykubat University
Organization: Alanya Alaaddin Keykubat University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: September 11, 2024 ID: 20-09
Record Dates: First submitted 2026-01-09; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Shock; Shock Circulatory
Keywords: Arterial blood gas; Emergency department; Radial artery puncture; Shock; Ultrasound
MeSH Terms: conditions — Shock; Emergencies

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized controlled trial. Patients were randomized in a 1:1 ratio into two groups using an online randomization tool. In the US group, arterial blood gas sampling was performed via radial artery puncture under real-time US guidance. In the non-US group, arterial blood gas sampling was performed using the conventional palpation technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Radial Artery Puncture (Experimental): Participants undergo radial artery puncture for arterial blood gas sampling using real-time ultrasound guidance.
  Interventions: Procedure: Ultrasound-guided radial arterial puncture for arterial blood gas sampling
- Conventional Palpation-Guided Radial Artery Puncture (Experimental): Participants undergo radial artery puncture for arterial blood gas sampling using the conventional palpation technique, which represents the standard practice.
  Interventions: Procedure: Conventional radial artery puncture for arterial blood gas sampling

INTERVENTIONS:
Procedure: Ultrasound-guided radial arterial puncture for arterial blood gas sampling — Radial artery puncture for arterial blood gas sampling performed under real-time ultrasound guidance. The artery is visualized on the screen and the needle is advanced under direct visualization until arterial blood flow is obtained.
  Arms: Ultrasound-Guided Radial Artery Puncture
Procedure: Conventional radial artery puncture for arterial blood gas sampling — Radial artery puncture for arterial blood gas sampling performed using the conventional palpation technique. The artery is identified by manual palpation and the needle is advanced until arterial blood flow is obtained.
  Arms: Conventional Palpation-Guided Radial Artery Puncture

SUMMARY:
Doctors in the emergency department often need to take blood samples from an artery to understand how well a patient is breathing and how the body is responding to serious illness. This is usually done by inserting a needle into an artery at the wrist. In patients with shock, this procedure can be difficult because blood pressure is low and the pulse may be hard to feel.

In this study, two different methods for obtaining arterial blood samples were compared in adult patients presenting to the emergency department with shock. In one group, the radial artery puncture was performed with ultrasound guidance, allowing direct visualization of the artery. In the other group, the procedure was carried out using the conventional palpation technique based on manual detection of the pulse.

Patients were randomly assigned to one of the two techniques. The study assessed the success of the procedure on the first attempt, the total number of attempts required, the time needed to obtain a successful sample, and whether puncture of the femoral artery was required when radial access could not be achieved.

The aim of the study was to evaluate whether the use of ultrasound improves the efficiency and success of radial artery blood sampling in patients with shock treated in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients diagnosed with shock
* Patients with an indication for arterial blood gas analysis due to respiratory or metabolic disorders
* Patients who provided written informed consent, either personally or through their legal representatives.

Exclusion Criteria:

* Patients who declined to participate
* Patients presenting with cardiac arrest
* Patients with a positive Allen test
* Patients with a history of coagulopathy
* Patients with evidence of infection at the puncture site
* Patients with evidence of trauma at the puncture site
* Patients with an arteriovenous fistula at the puncture site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
First-Attempt Success of Radial Artery Puncture | During procedure
  In the ultrasound-guided group, a stopwatch was started when the ultrasound transducer made contact with the skin over the radial artery. The artery was visualized on the screen, and the needle was advanced under real-time ultrasound guidance until arterial blood flow was obtained. The stopwatch was stopped when arterial blood flow was observed in the syringe, and the procedure was considered successful. Each new puncture attempt was recorded as a separate attempt.
  In the conventional palpation group, a stopwatch was started when the physician made skin contact after identifying the radial artery by palpation. The needle was advanced into the radial artery until arterial blood flow was obtained. The stopwatch was stopped when arterial blood flow was observed in the syringe, and the procedure was considered successful. Each new puncture attempt was recorded as a separate attempt.

SECONDARY OUTCOMES:
The Number of Attempts | During procedure
  Secondary outcomes included the number of attempts until successful puncture, time to successful puncture, and the need for a rescue femoral artery puncture.

OTHER OUTCOMES:
Procedure-Related Complications | within the emergency department stay (up to 4 hours after procedure)
  Occurrence of any procedure-related complications during or following radial artery puncture.

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Alaaddin Keykubat University Hospital, Alanya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data related to the primary and secondary outcomes will be shared upon reasonable request to the corresponding author.
Supporting Information: Study Protocol, SAP